CLINICAL TRIAL: NCT05096572
Title: A Randomized Cross-Over Trial of Deep Brain Stimulation (DBS) of the Posterior Subthalamic Area (PSA), Ventral Intermediate Nucleus of the Thalamus (VIM), and VIM+PSA on Essential Tremor (ET)
Brief Title: DBS of Posterior Subthalamic Area (PSA) and Ventral Intermediate Nucleus (VIM) in Essential Tremor (ET)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of enrollment
Sponsor: St. Joseph's Hospital and Medical Center, Phoenix (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 21-500-225-80-04
Record Dates: First submitted 2021-10-25; First posted 2021-10-27 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Essential Tremor
MeSH Terms: conditions — Essential Tremor

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (3):
- Group 1 (Experimental): Subjects will receive VIM stimulation for two weeks, followed by VIM+PSA stimulation for two weeks, and finally PSA stimulation for two weeks.
  Interventions: Device: VIM Stimulation; Device: PSA Stimulation; Device: VIM+PSA Stimulation
- Group 2 (Experimental): Subjects will receive VIM+PSA stimulation for two weeks, followed by PSA stimulation for two weeks, and finally VIM stimulation for two weeks.
  Interventions: Device: VIM Stimulation; Device: PSA Stimulation; Device: VIM+PSA Stimulation
- Group 3 (Experimental): Subjects will receive PSA stimulation for two weeks, followed by VIM stimulation for two weeks, and finally VIM+PSA stimulation for two weeks.
  Interventions: Device: VIM Stimulation; Device: PSA Stimulation; Device: VIM+PSA Stimulation

INTERVENTIONS:
Device: VIM Stimulation — Subjects will receive stimulation at VIM site only based on best settings ascertained during monopolar review.
Device: PSA Stimulation — Subjects will receive stimulation at PSA site only based on best settings ascertained during monopolar review.
Device: VIM+PSA Stimulation — Subjects will receive stimulation at VIM+PSA based on best settings ascertained during monopolar review.

SUMMARY:
Deep brain stimulation (DBS) of the ventral intermediate nucleus of the thalamus (VIM) is an FDA approved treatment for medication refractory essential tremor (ET). However, VIM stimulation can be associated with impacts on speech and balance. There is also suggestion that there may be habituation to stimulation in more than half of these patients. Stimulation of the posterior subthalamic area (PSA) has been found to be beneficial in tremor control as well. In fact, there is thought that the improvement in tremor in standard VIM DBS stimulation may be related to stimulation effects on the PSA. Updates in DBS stimulation allow to stimulate more than one area of the brain independently, while using a single lead. In this study, we will recruit patient who are referred for VIM DBS to a randomized cross-over trial in which they will receive VIM, PSA, or dual stimulation. We will assess tremor qualitatively and quantitatively, in addition to evaluating side effects, including quantitative gait analysis on each setting. The pre-operative, operative, and initial programming evaluation will be performed per standard of care. After baseline assessment and initial programming, subjects will be evaluated in a blinded manner after they have been on each setting for 2 weeks. The entire duration of the study from baseline visit through final study visit will be 17 weeks. For subjects who are clinically evaluated in our outpatient clinics, we will review their charts at 6 months for stimulation parameters and clinical information as it relates to their tremor.

DETAILED DESCRIPTION:
Essential Tremor (ET) is the most common movement disorder. It is estimated that between 25 and 55% of patients with ET will have a tremor which is refractory to pharmacotherapy necessitating advanced therapeutic options to control tremor. Deep Brain Stimulation (DBS) is one such option and has been FDA approved for ET since 1997 with the ventral intermediate nucleus of the thalamus (VIM) as a target. Over the past twenty years, DBS has become the standard of care for patients with treatment-refractory motor circuit disorders such as Parkinson's disease, dystonia, and essential tremor. A study reviewing the United States database hospital discharges from 2002 to 2011 showed that more than 30,000 DBS surgeries were performed during this time, 22% were for ET and the other 78% for Parkinson's Disease. A study done at Columbia University Medical Center estimated that about 1 in 34 ET patients undergo DBS surgery. DBS is highly effective at controlling motor symptoms and improvement in tremor with DBS in ET patients has been reported to be between 47.4% and 65.4%. However, there are limitations to stimulation in regard to adverse effects, such as dysarthria, gait imbalance, ataxia, etc. Additionally, some reviews suggest a loss of benefit in more than half, and as high as 73%, of individuals at a mean interval of approximately 18 months. Although DBS is relatively safe and effective, alternative surgical treatments include lesional therapies such as radiofrequency ablation, radiosurgery, and magnetic-resonance-guided focused ultrasonography. DBS still remains the standard of choice given ability to adjust stimulation over time or to turn it off if needed.

In addition to the VIM, the posterior subthalamic area (PSA) has emerged as a potential alternative target for ET. The PSA contains the Zona incerta (Zi) and prelemniscal radiation (Raprl) and has previously been targeted in subthalamotomies for tremor control. It is believed that the cerebellothalamic connections of the PSA are involved in tremor and that the somatotopic organization of the PSA allows for improvement in proximal tremor control, in particular. From a stimulation perspective, results published in the literature have suggested that the PSA may be equivalent, and possibly superior to the VIM, in terms of therapeutic benefit. The PSA was targeted in a case series of patients with severe proximal tremor specifically, and found to have beneficial impact. The VIM is located dorsal to the PSA which allows for access to both structures with a single electrode and in fact, review of VIM lead locations and optimal contacts for tremor control have shown better tremor control with more ventral contacts, which are more likely stimulating the PSA, to have superior tremor control than that achieved with thalamic stimulation.

A single small study evaluated the surgical approach of targeting both VIM and PSA with a single electrode for dual stimulation and found this to be a feasible surgical procedure. This study showed equivalent outcomes for VIM, PSA, and VIM+PSA but this was a small unblinded study with only 8 patients. Another small study assessing 17 patients with ET and DBS of both VIM and PSA in one surgical trajectory found that intraoperatively, PSA stimulation offered superior tremor control compared to VIM in 88% of aligned trajectories. Dysarthria and gait ataxia were side effects seen in both VIM and PSA stimulation. Successful tremor control was achieved in 69% of patients.

In our center, we have a series of patients with longstanding ET who initially had considerable improvement of tremor following DBS of the VIM only. Although this benefit was sustained for several years, these patients had re-emergence of their tremor requiring increasing stimulation over time as well as reintroduction of pharmacotherapy for tremor control. Higher stimulation was limited by adverse effects in the form of dysarthria and ataxia. Given the significant disability from their tremors, and the availability of newer DBS leads with more contacts and the availability of complex stimulation options, these individuals underwent replacement of their existing VIM DBS leads with longer leads targeting both the VIM and PSA in one surgical trajectory as salvage therapy. Retrospective review of these cases show that the reduction in tremor was higher for those receiving concurrent VIM and PSA stimulation compared to VIM or PSA alone. Others had a reduction in their tremor but were still functionally limited as even with considerable reduction in tremor amplitude, there was still a robust tremor present. However, this is a small case series of severely refractory ET and broad generalizations cannot be made. Therefore, we propose a prospective, randomized, cross-over trial of DBS for ET quantitatively assessing whether dual stimulation of VIM and PSA is superior to VIM or PSA alone in terms of the various tremor components of ET (i.e. proximal v. distal limb tremor), quality of life measures, and side effect profile. We postulate that since two targets involved in tremor control will be stimulated simultaneously, lower current will be needed at each target which should limit involvement of adjacent pathways which are typically recruited with higher stimulation and lead to side effects.

This study will not be an evaluation of a new surgical target or trajectory, as the patients eligible to be recruited for this study will already be candidates for VIM+PSA DBS, which are closely positioned and connected structures often affected simultaneously by DBS depending on lead placement and targeting of stimulation. This study will only be examining the separate and combined affected of stimulation within these two structures using the more accurate targeting available with GuideXT software.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with a diagnosis of ET, refractory to pharmacotherapy referred for DBS consideration.
* Informed consent signed by the subject.
* DBS candidate per FDA guidelines.
* Primary language - English
* Physically and cognitively capable of completing evaluations and consent
* Medically cleared for surgery and anesthesia
* Negative pregnancy test prior to surgery for female subjects of child-bearing potential.

Exclusion Criteria:

* Any individuals with contraindication to bilateral DBS lead placement, history of dementia per DSM-V criteria, intracranial hemorrhage, or psychiatric illness.
* Conditions precluding MRI.
* History of supraspinal disease.
* Subjects with a history of seizure disorder.
* Subjects who have made a suicide attempt within the prior year,
* Subjects with any medical contraindications to undergoing DBS surgery (eg, infection, coagulopathy, or significant cardiac or other medical risk factors for surgery)
* Subjects with an implanted stimulator such as a cardiac pacemaker, defibrillator, neurostimulator and cochlear implant
* Subjects who are pregnant or nursing.
* Patient that is unwilling or unable to comply with the requirements of this protocol, including the presence of any condition (physical, mental, or social) that is likely to affect the subject's ability to comply with the protocol.
* Any other reasons that, in the opinion of the investigator, the candidate is determined to be unsuitable for entry into the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2021-11-30 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2023-10-30 (Actual)

PRIMARY OUTCOMES:
Improvement in Tremor | Following Two Weeks of Treatment At Each Intervention
  Tremor will be measured quantitatively using inertial measurement units. FTM-TRS will also be measured by the investigator.
Change in Tremor Phenomenology | Following Two Weeks of Treatment At Each Intervention
  Frequency and amplitude will be measured quantitatively using IMUs during postual, action, and intentional tasks.
Change in Stimulation-Induced Balance | Following Two Weeks of Treatment At Each Intervention
  Quantitative gait assessment utilizing the Zeno Walkway System will measure changes in balance at each visit.
Change in Stimulation-Induced Dysarthria | Following Two Weeks of Treatment At Each Intervention
  A dysarthria visual analog scale will measure dysarthria.

CONTACTS AND LOCATIONS:
Overall Officials: Sana Aslam, DO, Principal Investigator — St Josephs Hospital and Medical Center
Locations (1):
- Barrow Neurological Institite, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No